CLINICAL TRIAL: NCT04314609
Title: The Success Rate of Ultrasound Guided Sacroiliac Joint Steroid Injections in Sacroiliitis: Are we Getting Better
Brief Title: Success Rate of Ultrasound Guided Sacroiliac Joint Injection in Sacroiliitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karim Alaaeldin Tawfik (Other)
Responsible Party: Sponsor-Investigator, Karim Alaaeldin Tawfik, Doctor, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-161-2018
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Sacroiliitis
MeSH Terms: conditions — Sacroiliitis | interventions — Ultrasonography; Fluoroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound , fluroscope (Experimental): After injection of corticosteroids with 1 ml contrast in sacroiliac joint using ultrasound and withdrawal of the needle, an antero-posterior fluoroscopy image will be obtained and recorded for the injected joint to detect the spread pattern of the contrast and whether its pre-dominantly intra or periarticular.
  Interventions: Device: Ultrasonography, fluoroscopy

INTERVENTIONS:
Device: Ultrasonography, fluoroscopy — success rate of Ultrasound guided SIJ steroid injection confirmed by contrast spread in fluoroscopy

SUMMARY:
To re-investigate the success rate of Ultrasound guided sacroiliac joint steroid injection in depositing the drug inside the joint capsule (confirmed by contrast spread in fluoroscopy) and if there is a difference in clinical outcome between injections done strictly inside the joint and injections done periarticular.

DETAILED DESCRIPTION:
An IV cannula will be inserted, and basic ASA monitors applied, then the patients will be positioned in prone position. After disinfection of the skin, Ultra sonography will be used to Guide Needle Placement in SIJ (the hypoechoic cleft between the surface of the sacrum and the ilium) under complete a sepsis as the technique previously described in the literature.

A low frequency (2-5 Hz) curvilinear transducer will be used in a sterile cover, the posterior superior iliac spine, lateral borderof sacrum, and ilium will be identified in transverse orientation. Subsequently, the probe will be moved caudally until the superior part of the posterior SIJ is identified. The SIJ will be traced caudally until the distal third of the SIJ is visualized as evident by the flat contour of the iliac crest and the presence of the second sacral foramen on the medial aspect of the sacrum.

After local anesthetic infiltration of skin and subcutaneous tissues using Lidocaine 1%, a 21-gauge spinal needle will be advanced from a medial to lateral direction using an in-plane technique. After reaching the joint, a total volume of 4 ml of injectate will be injected which consists of: 1 ml 40 mg of methylprednisoloneacetate (Depo-Medrol®, Pfizer), 2 ml Lidocaine 2%, 1 ml Iohexol (Omnipaque 300®, GE Healthcare).

Control fluoroscopy

After injection of the drug and withdrawal of the needle, a antero-posterior fluoroscopy image will be obtained and recorded for the injected joint to detect the spread pattern of the contrast and whether its pre-dominantly intra or periarticular. (N.B: Periarticular injection is any injection done near the joint as evidenced by US but on fluoroscopy no contrast is detected inside the joint). Then a sterile patch will be applied to the puncture site and patient discharged to the recovery room for follow-up for 30 minutes before discharge to home.

Measurement tools

* Total number of intraarticular and periarticular drug injections as evidenced by contrast spread in fluoroscopy.
* Patient's pain score rated from 0-10 (Numeric Pain Rating Scale, NRS) before the procedure, 10 minutes after the procedure (in the recovery room), 1 week and 1 month post-procedure.
* Demographic data (including age, sex, BMI, ASA score).
* Limitation of physical functioning as measured by the Oswestry Disability Index (ODI) at 1 month after the procedure .
* Procedure-related variables (time, complications, patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Subject has sacroiliitis (acute or chronic) by history.
* Failed conservative therapy eg. bed rest, anti-inflammatory medications and physical therapy for at least 6 weeks.

Exclusion Criteria:

* Subject has BMI above 35 kg/m2
* Coagulopathy.
* Renal or Hepatic Failure.
* Current Pregnancy or actively pursuing pregnancy.
* Known allergy to local anesthetic or steroids.
* Infection at site of needle placement or SIJ infection.
* Prior surgical procedures involving the SIJ.
* Previous surgical Fixation involving the lumbar spine.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
success rate of ultrasound sacroiliac joint injection | Immediately after injection
  Percent of successful intraarticular drug injections during USG SIJ steroid injection (as confirmed by contrast spread in fluoroscopy)

SECONDARY OUTCOMES:
Difference in clinical outcome between intraarticular and periarticular injections. | After 10 minutes, 1 week and 1 month
  Difference in clinical outcome between intraarticular and periarticular injections (confirmed via fluroscopy) as measured clinically by numerical pain score (NPS is a scale from 0 to 10. 0 is no pain and 10 is the maximum pain)
Clinical improvement | After 10 minutes, 1 week ,1 month
  Pain score at 10 minutes , 1 week and 1 month after intervention by numerical pain score (NPS is a scale from 0 to 10. 0 is no pain and 10 is the maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Amany E Ayad, M.D, Principal Investigator — Cairo University; Ahmed Z Fouad, M.D, Study Chair — Cairo University; Mohamed A Mansour, M.D, Study Chair — Cairo University; Karim A Tawfik, MSc, Study Chair — Cairo University
Locations (1):
- Faculty of medicine cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No